CLINICAL TRIAL: NCT04774302
Title: Study of Correlation Between Hepatic Fibrosis and Cardiovascular Risk Evaluated by Non-invasive Tests in Patients With Nonalcoholic Fatty Liver Disease
Brief Title: Correlation Between Hepatic Fibrosis and Cardiovascular Risk Evaluated by Non-invasive Tests in Patients With NAFLD
Acronym: Cardio-NASH
Status: Completed | Type: Observational
Sponsor: Clinique Pasteur (Other)
Responsible Party: Principal Investigator, Dr Maeva GUILLAUME, Principal investigator, MD, Clinique Pasteur
Other Study IDs: 2020-A03423-36
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: NAFLD
Keywords: CAC score; Liver fibrosis; Cardiovascular risk; Metabolic syndrome
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to examine the link between Non-Alcoholic Fatty Liver Disease (NAFLD) and cardiovascular diseases by studying the association between liver fibrosis degree and cardiovascular risk factors. The study would clarify the value and the role of the Coronary calcium score (CAC score) in the screening for coronary disease in this population at high cardiovascular risk.

DETAILED DESCRIPTION:
Hepatic Fibrosis and Cardiovascular Risk are evaluated by non invasive tests

ELIGIBILITY:
Inclusion Criteria:

* NAFLD patients regardless of disease stage of severity (from simple steatosis to cirrhosis)
* Patient without known heart disease
* Patient agreeing to participate and who has given his non opposition

Exclusion Criteria:

* Association with another cause of liver disease
* Already known coronary artery disease
* Pregnancy or breastfeeding in progress

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female evaluated in a dedicated hepatology day hospital, as part of a first diagnostic workup or follow-up for already known NAFLD
Sampling Method: Non-Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Coronary calcium score | At inclusion
  Score in Agatston IU of coronary atherosclerosis risk;ranging from 0 to 100 : low risk; 100 to 400 : intermediate risk and > 400 : high risk of coronary atherosclerosis.
Shear wave liver elastography | At inclusion
  Hepatic elasticity assessed in kPa : <5 Kpa : normal; 5 to 8 kPa : low to moderate fibrosis ; > 8 kPa : advanced fibrosis; >15 kPa : cirrhosis

SECONDARY OUTCOMES:
ARFI Hepatic elasticity | At inclusion
  Hepatic elasticity assessed by Acoustic radiation force impulse (ARFI) (in kPa) Hepatic elasticity assessed in kPa : <5 Kpa : normal; 5 to 8 kPa : low to moderate fibrosis ; > 8 kPa : advanced fibrosis; >15 kPa : cirrhosis .
Cardiovascular risk | At inclusion
  Systemic Coronary Risk Estimation (SCORE) ranging from <1% very low risk to >15% very high risk of cardiovascular mortality
Coronary heart disease | 3 month
  Diagnosis of coronary heart disease

CONTACTS AND LOCATIONS:
Overall Officials: Maeva GUILLAUME, MD, Principal Investigator — Clinique Pasteur
Locations (1):
- Clinique Pasteur, Toulouse, France